CLINICAL TRIAL: NCT04017273
Title: Older Emergency Department Users and Hospitalization After an Index Visit: Results of ER2 Database
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1882
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Chronic Conditions, Multiple; Medical Emergencies
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: The participants of this study will be seen at Emergency Department, and a nurse will perform a test called ER2 ( Emergency Room Evaluation and Recommendation).

SUMMARY:
This study evaluates the recommendations of a screening tool called: ER2 (Emergency Room Evaluation and Recommendations Form).This stool is used in Emergency Department by nurses, and it supposes to measure patient risk score.

DETAILED DESCRIPTION:
Crowding and delay became chronic conditions in emergency departments (EDs) in high income countries. Emergency medicine has the mandate to provide care to any patient requesting treatment 24 hours a day. As there is a lack of primary care physicians who are able to provide the necessary care to patients, they are forced to seek care in ED. Among these ED users, more and more patients are aged over 65 and account for up to a quarter of all ED users. Older ED users comparted to their younger counterparts are more at risk for long length of stay in ED and hospital, and hospital admission during an index ED visit. The occurrence of these short-terms adverse events may be reduced if older ED users risk is assessed upon their ED arrival. Few studies have examined risk for short-terms adverse events. They suggested that clinical tools based on a brief geriatric assessment with timely appropriate interventions could reduce the occurrence of short-terms ED adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Being 75 years and over
* Brought at Emergency on medical stretcher

Exclusion Criteria:

* Being less than 75 years old
* Never come at Emergency

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In this study will be enrolled people who are 75 years and over, and who come at Emergency not only for medical reason but also for social.
Sampling Method: Non-Probability Sample
Enrollment: 10971 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Long length of hospital stay | Around 10 months
  Long length of hospital stay represents an indicator of efficiency, and it refers to the average number of day that a patient spends in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada